CLINICAL TRIAL: NCT03678168
Title: A Comparison Between Conventional Throat Packs and Pharyngeal Placement of Tampons in Rhinology Surgeries
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Hamad University Hospital, Bahrain (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KHUH/216
Record Dates: First submitted 2018-08-19; First posted 2018-09-19 (Actual); Last update posted 2019-10-22 (Actual); Status verified 2019-10

CONDITIONS: Pain; Postoperative Pain; Bleeding; Nose Bleed
MeSH Terms: conditions — Pain; Pain, Postoperative; Hemorrhage; Epistaxis | interventions — Methods

STUDY DESIGN:
Who Masked: Participant
Masking Description: The participants will be unaware of the type of packaging used port rhinology surgery to control pain and bleeding.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control (Other): Standard care (Throat pack) which will be used as a control.
  Interventions: Other: Throat Pack
- Intervention (Experimental): Pharyngeal tampons which will be used as a comparator against throat pack.
  Interventions: Other: Pharyngeal Tampons

INTERVENTIONS:
Other: Throat Pack — Post rhinology surgery throat packs will be used as a control to compare against the intervention (Pharyngeal tampons)
  Other Names: Control
  Arms: Control
Other: Pharyngeal Tampons — Post rhinology surgery Pharyngeal Tampons will be used as an intervention to compare against the throat pack (control)
  Other Names: Intervention
  Arms: Intervention

SUMMARY:
Post-operative, throat pain, nausea and vomiting is a common occurrence in rhinology surgeries due to the use of throat packs during the procedure. In order to optimize quality of care and patient satisfaction, the aim of this study to evaluate the incidence of post-operative, throat pain, nausea and vomiting in patients that have been packed with either conventional gauze throat packs or pharyngeal tampons.

DETAILED DESCRIPTION:
The nose and para nasal sinuses are anatomically known to be highly vascular and a substantial amount of bleeding is expected from rhinology surgeries, ingested blood is known to be a power full emetic, and the risk aspiration of blood is present due to the fact that an endotracheal tube is not 100% effective in protecting the airway. Post-operative nausea and vomiting is a frequent problem that is encountered in surgical patients with a 4th to 6th fold increase in nasal and endoscopic sinus operations.

Posterior throat pack is an often-used in rhinology surgery, it is said to help in protecting the air way against aspiration and also helps in the reduction of post-operative nausea and vomiting, however many studies concluded that posterior throat pack is associated with higher amount of post-operative pain, nausea,, vomiting and in some rare cases even forgotten in the patient leading to mortality. However, despite poor evidence the placement of posterior throat packs is commonly practiced by surgeons and anesthetists because the possible risk of aspiration is worrisome to the latter and the former.

A conventional throat pack consists of gauze, but an alternative practice involves the pharyngeal placement of tampons. In Marais and Prescott posterior pharyngeal placement of tampons is associated with a decrease amount of post-operative throat pain, when compared to conventional gauze throat packs, however they did not compare the incidence of post-operative nausea and vomiting in both groups.

ELIGIBILITY:
Inclusion Criteria:

* Adults patients ( above the age of 18 years)
* Admitted under Dr. Hiba Al-Reefy
* Underwent a rhinology procedure that required the use of a throat pack

Exclusion Criteria:

* Pediatric patients
* Pt who underwent a procedure without the use of throat packs

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 86 (Actual)
Dates: Start 2018-09-05 (Actual); Primary Completion 2019-08-15 (Actual); Study Completion 2019-09-15 (Actual)

PRIMARY OUTCOMES:
Comparison of postoperative throat pain using the visual analogue scale (VAS) | 2 years
  Evaluation of postoperative pain between pharyngeal tampons and controls using the Visual Analogue scale. A value of 0 is the lowest value and indicates the patient is pain free. And a score of 10 is the maximum value which indicates extreme pain on the scale.
postoperative throat bleed | 2 years
  Evaluation of postoperative bleeding in patients using pharyngeal tampons vs control

SECONDARY OUTCOMES:
Postoperative recovery | 2 years
  Assess the postoperative symptom recovery

CONTACTS AND LOCATIONS:
Locations (1):
- King Hamad University Hospital, Al Muharraq, Muharraq, Bahrain, Bahrain

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Piltcher O, Lavinsky M, Lavinsky J, de Oliveira Basso PR. Effectiveness of hypopharyngeal packing during nasal and sinus surgery in the prevention of PONV. Otolaryngol Head Neck Surg. 2007 Oct;137(4):552-4. doi: 10.1016/j.otohns.2007.04.004. PMID 17903569
- [Background] Fennessy BG, Mannion S, Kinsella JB, O'Sullivan P. The benefits of hypopharyngeal packing in nasal surgery: a pilot study. Ir J Med Sci. 2011 Mar;180(1):181-3. doi: 10.1007/s11845-010-0601-4. Epub 2010 Nov 26. PMID 21110138
- [Background] Seraj MA, Ankutse MM, Khan FM, Siddiqui N, Ziko AO. Tracheal soiling with blood during intranasal surgery--comparison of two endotracheal tubes. Middle East J Anaesthesiol. 1991 Feb;11(1):79-89. PMID 2067508
- [Background] Jaiswal V, Bedford GC. Review of the use of throat packs in nasal surgery. J Laryngol Otol. 2009 Jul;123(7):701-4. doi: 10.1017/S0022215109004356. Epub 2009 Feb 4. PMID 19192316
- [Background] Tay JY, Tan WK, Chen FG, Koh KF, Ho V. Postoperative sore throat after routine oral surgery: influence of the presence of a pharyngeal pack. Br J Oral Maxillofac Surg. 2002 Feb;40(1):60-3. doi: 10.1054/bjom.2001.0753. PMID 11883973